CLINICAL TRIAL: NCT05753787
Title: Assessment of the Eye Surface and Subjective Symptoms After Using Dexamethasone Drops With and Without Preservatives in Patients After Cataract Surgery
Brief Title: Eye Surface Properties After Using Dexamethasone Drops With and Without Preservatives in Patients After Cataract Surgery
Acronym: EyeSurface
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spektrum Center of Clinical Ophthalmology (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Spektrum2022/01
Record Dates: First submitted 2022-10-23; First posted 2023-03-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cataract; Surgical Injury; Healing Wound
MeSH Terms: conditions — Cataract; Intraoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preservatives-free dexamethasone 0.1% eye drops (Active Comparator)
  Interventions: Other: preservative-free solution of standard post-cataract eye drops
- preserved dexamethasone 0.1% eye drops (Placebo Comparator)
  Interventions: Other: preservative-free solution of standard post-cataract eye drops

INTERVENTIONS:
Other: preservative-free solution of standard post-cataract eye drops — Usage of preservative-free eye drops in comparison to the standard preserved drops with dexamethasone 0.01%.

SUMMARY:
The goal of this interventional, real world data study is to evaluate the impact of preservatives on the post-cataract ocular surface.

The main question is to learn about an effect of preservatives on the eye surface. The study aims to answer some important questions:

* if the usage of preservatives has an impact on the eye surface healing process after cataract surgery
* if patient comfort and quality of life improve more or more rapidly with preservatives-free eye drops.

Participants will be asked to undergo standard procedure of peri-cataract surgery care and in addition to survey about the ocular surface state.

Researchers will compare group that takes preservatives-free dexamethasone 0.1% with standard dexamethasone 0.01% solution to see if post-surgery eye surface healing properties differ from both groups.

ELIGIBILITY:
Inclusion Criteria:

* cataract surgery required defined previously by the eye-care specialist
* good and clear visibility of the anterior chamber in the pre-surgery status (enables investigators to assess the anterior chamber cell intensity)
* consent to the study protocol

Exclusion Criteria:

* diagnosed glaucoma
* diagnosed previous allergy
* diagnosed diabetic retinopathy or maculopathy
* previously diagnosed dry eye disease that requires treatment with multiple artificial tears
* permanent usage of the eye drops other than artificial tears
* non-compliance to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity result | up to 21 days post-surgery
  best corrected visual acuity evaluated with standard ETDRS for distant and for near vision
Ocular staining score result | up to 21 days post-surgery
  standard staining score - a scale used with the fluorescein stain; higher value expres more severe outcome, normal values are around 0-1. Overal information can be found: https://entokey.com/a-simplified-quantitative-method-for-assessing-keratoconjunctivitis-sicca-from-the-sjogrens-syndrome-international-registry/
Ocular Surface Disease Index survey result | up to 21 days post-surgery
  a standard survey that patient will preform at each visit

SECONDARY OUTCOMES:
Fluorescein Break-up Time assessment | up to 21 days post-surgery
  time to break-up the tear film after the instilation of the fluorescein eye drop (evaluated 3 fold and the mean will be taken into account)
SICCA scale assessment | up to 21 days post-surgery
  Scale that requires both fluorescein and lissamine green staining profile assesment - used in the standardised manner
Shirmer test 1 measurement | up to 21 days post-surgery
  test that evaluate the amount of tears (in mm on the test paper) that are produced within 5 minutes and are evaluated under the anesthesia
Intraocular pressure measurement | up to 21 days post-surgery
  Intraocular pressure measurement preformed by standard tonometer
Anterior chamber cell intensity measurement | up to 21 days post-surgery
  the standardised SUN assesment of the anterior chamber cell intensity will be preformed - a standardised scale

CONTACTS AND LOCATIONS:
Overall Officials: Maria Muzyka-Woźniak, PhD, Principal Investigator — Spektrum Clinic of Ophthalmology
Locations (1):
- Spektrum Clinic of Ophthalmology, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muzyka-Wozniak M, Strozecki L, Przezdziecka-Dolyk J. Assessment of the eye surface and subjective symptoms after using 0.1% dexamethasone drops with and without preservatives in patients after cataract surgery. Sci Rep. 2023 Oct 30;13(1):18625. doi: 10.1038/s41598-023-44939-1. PMID 37903818